CLINICAL TRIAL: NCT01727310
Title: Filling Pressures of the Left Ventricle in Patients With Significant Aortic Stenosis: Study of Echocardiographic Parameters Compared to Invasive Evaluation
Brief Title: Filling Pressures of the Left Ventricle in Patients With Significant Aortic Stenosis
Acronym: PRESSEVAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I10013
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Valvular Disease

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Left valvular heart disease has become one of the most common heart disease in Western countries. This disease evolve over many years and are characterized by a long phase where the patient is "asymptomatic".

it is characterized by discomfort LV filling may worsen and lead typically to a pressure increase of LV pressure and the left atrium (LA) (1). The onset of symptoms is unpredictable and may occur at the stage of diastolic or systolic dysfunction.

Ventricular dysfunction may be insidious, the goal is to detect early dysfunction, knowing that it is often very difficult to know if the patient is actually symptomatic. The onset of symptoms sign an intolerance to the increase in LV filling pressures and LA , causing pulmonary hypertension .

Therefore, the study of the level of LV and LA filling pressures , if possible by a noninvasive method, would identify patients apparently asymptomatic even though their condition is advanced.

Pressures filling pressures can be explored by two methods:

* cardiac catheterization, which is a direct and invasive measurement method
* echocardiography, which is an indirect measurement method which has the advantage of being non-invasive The goal of this research is to compare the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years;
* Patients hospitalized for a coarctation review, and has received or will be receiving during their stay a complete echocardiography and coronary angiography, and left and right catheterization

Exclusion Criteria:

* Pregnant women
* Patients with a history of valve replacement surgery,
* Patients with other valvular> grade 2 associated with the coarctation
* Patients known to have ischemic heart disease or in whom angiography showed significant coronary artery disease;
* Patients with chronic or paroxysmal atrial fibrillation
* Patients with a permanently pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both gender hospitalized for a coarctation review, and has received or will be receiving during their stay a complete echocardiography and coronary angiography, and left and right catheterization .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
quality of echocardiography
  Evaluate the diagnostic quality of echocardiography to measure the volume of the LA indexed to body surface area compared to cardiac catheterization

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Departement de Cardiologie, Limoges
  - Departement de Cardiologie, Montpellier